CLINICAL TRIAL: NCT05896592
Title: A Multicenter, Randomized, Double-blind, Research Study comparinG the Efficacy and Safety of cardioneuroablaTion vs Permanent Pacing in Patients With an implantabLE PACEmaker for Symptomatic Bradycardia.
Brief Title: Comparison of the Efficacy and Safety of Cardioneuroablation to Permanent Pacing in Patients With an Implanted Pacemaker for Symptomatic Bradycardia.
Acronym: GENTLE-PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4th Military Clinical Hospital with Polyclinic, Poland (Other)
Responsible Party: Principal Investigator, Przemysław Skoczyński, MD, PhD, 4th Military Clinical Hospital with Polyclinic, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/2023
Record Dates: First submitted 2023-05-21; First posted 2023-06-09 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Bradycardia; Syncope
Keywords: cardioneuroablarion; functional bradycardia; pacemaker treatment discontinuation
MeSH Terms: conditions — Bradycardia; Syncope | interventions — Electrocardiography, Ambulatory; Immunologic Memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The project is a double-blind study. Blinding will only apply to the study arms with group 1 and 2. Neither the researcher (doctor) nor the participant (patient) will know what invasive procedures will be performed on a given patient. Patients, investigators, and everyone involved in conducting or analyzing the study, along with other persons interested in the results of the study, will remain blinded to the treatment assigned to individual patients (CNA with continuation of PM therapy vs. continuation of PM therapy without CNA) from the beginning of the study until the database is closed. The operator performing EPS, ECVS, CNA and ILR implantation will not be blinded. Operator will not be involved in the subsequent management of the patient in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 will undergo EPS, ECVS, CNA with continuation of PM therapy and ILR implantation. Two months later pacing rate, will be assessed. In addition, there will be a non-invasive assessment of the effectiveness of CNA. After another month, EPS and ECVS will be performed and a re-CNA if the ECVS does not show full parasympathetic denervation of the heart. The pacemaker will be set to VVI or AAI 30/min. One month after the second invasive procedure, the pacing rate will be assessed. Patients with zero percentage of PM stimulation will be set to ODO/OVO/OAO-stimulation off mode. Patients will be monitored for the next 12 months. During the next 4 visits repeated every 3 months, patients in this group will undergo non-invasive assessment of the effectiveness of CNA and symptoms of bradycardia. At the 7th visit, patients in this group will be qualified to discontinue of the cardiac pacing treatment, with possible qualification for TLE.
  Interventions: Diagnostic Test: Invasive electrophysiological study; Diagnostic Test: Extracardiac vagal stimulation; Procedure: Cardioneuroablation; Procedure: Redo cardioneuroablation; Procedure: Implantation of the implantable loop recorder; Diagnostic Test: Pacemaker check; Diagnostic Test: Implantable loop recorder check; Diagnostic Test: Holter ECG; Diagnostic Test: Anamnesis
- Group 2 (Experimental): Group 2 will undergo EPS and ECVS with continuation of PM therapy, ILR implantation, without CNA. Two months later pacing rate, will be assessed. After another month, EPS, ECVS and CNA will be made. The pacemaker will be set to VVI or AAI 30/min. One month after the second invasive procedure, patients in this group will have their pacing rate assessed. Patients with zero percentage of PM stimulation will be set to ODO/OVO/OAO-stimulation off mode. Patients will be monitored for the next 12 months. During next 4 visits repeated every 3 months, patients in this group will undergo a non-invasive assessment of the effectiveness of CNA and symptoms of bradycardia. At the 7th visit, the qualification for discontinuation of cardiac pacing treatment will take place, with possible qualification for TLE.
  Interventions: Diagnostic Test: Invasive electrophysiological study; Diagnostic Test: Extracardiac vagal stimulation; Procedure: Cardioneuroablation; Procedure: Implantation of the implantable loop recorder; Diagnostic Test: Pacemaker check; Diagnostic Test: Implantable loop recorder check; Diagnostic Test: Holter ECG; Diagnostic Test: Anamnesis
- Group 3 (Active Comparator): Group 3 patients will only be observed for the duration of the study. The observation period will be 18 months. At subsequent visits 1, 3, 4, 6, 9, 12, 15 months after randomization, they will be assessed for the presence of MAS, paraMAS and assessment of the percentage of stimulation.
  Interventions: Diagnostic Test: Pacemaker check; Diagnostic Test: Anamnesis

INTERVENTIONS:
Diagnostic Test: Invasive electrophysiological study — Invasive electrophysiological study consists in inserting two electrodes into the heart through femoral vein puncture into the right atrium and right ventricle. Then the following measurements are taken: SNRT- sinus rhythm recovery time, cSNRT- corrected sinus rhythm recovery time, Wenckebach point, AH and HV time and HRV-rhythm variability after SNRT measurement. The examination will be performed under general anesthesia.
  Other Names: EPS
  Arms: Group 1; Group 2
Diagnostic Test: Extracardiac vagal stimulation — Extracardiac vagal stimulation consists in leading the electrode through the puncture of the femoral vein, successively to both internal jugular veins and stimulating the vagus nerve at the level of its cranial orifice and lower at the level of the angle of the mandible. Stimulation is performed using the Extra-Cardiac Autonomic NeuroStimulatorPachon.
  Induction of a sinus pause or AV block during vagal stimulation is considered a positive test result. Absence of sinus pause and AV block during vagal stimulation indicates parasympathetic denervation of the heart. The examination is performed under general anesthesia.
  Other Names: ECVS
  Arms: Group 1; Group 2
Procedure: Cardioneuroablation — CNA consists in complete parasympathetic denervation of the heart or in its deep neuromodulation by destroying the postganglionic nerve fibers of the vagus nerve, located in the epicardium in the vicinity of the pulmonary veins to the left atrium and in the area of the interatrial septum. It consists in inserting the electrode into the left atrium through puncture of the femoral vein, and then the interatrial septum, and performing ablation in the vicinity of the pulmonary vein orifices and on the interatrial septum at the level of the mitral annulus. Then the electrode is withdrawn into the right atrium and subsequent applications are made in the area of the coronary sinus opening and the roof of the right atrium and the upper part of the interatrial septum. The procedure is performed under general anesthesia. In group 1, CNA will be performed 1 month after randomization. In group 2, CNA will be performed 4 months after randomization.
  Other Names: CNA
  Arms: Group 1; Group 2
Procedure: Redo cardioneuroablation — It consists in re-performing the CNA if full parasympathetic parasympathetic denervation of the heart is not confirmed by ECVS.
  Other Names: redo CNA
  Arms: Group 1
Procedure: Implantation of the implantable loop recorder — Implantation of the implantable loop recorder consists in subcutaneous implantation of the ECG loop recorder in the sternum area.
  Other Names: ILR implantation
  Arms: Group 1; Group 2
Diagnostic Test: Pacemaker check — It consists in evaluating the reliability of the PM system. And the assessment of pacing percentage and recorded arrhythmias. After successful cardioneuroablation in groups 1 and 2, 4 months after randomization, the PM will be programmed to the VVI 30/min mode and after 6 months to the OAO/OVO mode. In group 3 patients and in the case of unsuccessful cardioneuroablation, the pacemaker will be set to the optimal mode for the patient. During the PM control, a non-invasive electrophysiological study (NIEPS) is also performed, in which the SNRT, cSNRT, Wenckebach point and HRV after SNRT measurement are assessed. The procedure will be repeated at subsequent visits 1, 3, 4, 6, 9, 12, 15, 18 months after randomization.
  Other Names: PM check
Diagnostic Test: Implantable loop recorder check — Assessment of arrhythmias recorded in the ILR. The procedure will be repeated at subsequent visits 3, 4, 6, 9, 12, 15, 18 months after randomization.
  Other Names: ILR check
  Arms: Group 1; Group 2
Diagnostic Test: Holter ECG — 24 hour ECG recording. The procedure will be repeated at subsequent visits 1, 3, 4, 6, 9, 12, 15, 18 months after randomization.
  Arms: Group 1; Group 2
Diagnostic Test: Anamnesis — Medical history assessing symptoms of bradycardia, MAS, paraMAS and complications of performed procedures. The procedure will be repeated at subsequent visits 1, 3, 4, 6, 9, 12, 15, 18 months after randomization.

SUMMARY:
Background Sinus node dysfunction (SND) and atrioventricular block (AVB) are significant diagnostic and therapeutic problems. The primary method of their treatment is cardiac pacemaker implantation (PM). Although PM remains the main therapeutic approach for most patients with SND/AVB, long-term PM therapy can be associated with various limitations, complications, and the need for device and electrode replacement. There is increasing evidence for the effectiveness of an alternative approach to functional bradycardia associated with excessive vagal activation - cardioneuroablation (CNA). The method leads to the alleviation or complete resolution of bradycardia symptoms, as well as reflex syncope, providing an opportunity to discontinue PM therapy.

Primary aims

1.Evaluation of the efficacy and safety of CNA as a therapy allowing for discontinuation of PM therapy in patients with SND or AVB.

Secondary aims

1. Evaluation of the efficacy and safety of CNA as a therapy allowing for the optimization of PM therapy in patients with SND and AVB.
2. Development of a diagnostic algorithm allowing for the identification of patients with SND and/or AVB suitable for CNA and discontinuation of PM and TLE therapy.
3. In addition, blood samples will be collected for future analysis and biobanking.

Methodology

Inclusion criteria

1. Patients up to 50 years old who underwent pacemaker implantation due to sinus node and/or atrioventricular node dysfunction
2. Positive response to atropine test
3. Age between 18-65 years
4. Signed informed consent to participate in the study

Exclusion criteria

1. Own heart rate <30/min
2. Fainting after pacemaker therapy initiation
3. Persistent and sustained atrial fibrillation
4. History of myocarditis
5. History of myocardial infarction
6. History of cardiac surgery
7. History of ablation procedures
8. Congenital heart defects
9. Congenital atrioventricular block
10. Neuromuscular and neurodegenerative diseases
11. Indications for expanding the pacemaker system to ICD/CRT-D
12. Pregnancy
13. Renal insufficiency with GFR <30 ml/min/1.73m2
14. Age below 18 and above 65 years
15. HAS-BLED score >/= 3 points

Randomization, study scheme Qualified patients will be randomly assigned (1:1:1) to group 1 undergoing first-stage invasive electrophysiology study (EPS), extracardiac vagus nerve stimulation (ECVS) and CNA with continued PM therapy and implantable loop recorder (ILR) implantation, to group 2 undergoing first-stage EPS and ECVS with continued PM therapy, ILR implantation, and no CNA, and to group 3 where patients will undergo observation only for the entire study. The follow-up time will be 18 months. Groups 1 and 2 will be blinded. Two months after the first invasive procedure, the secondary endpoint-stimulation rate in all groups will be assessed. In addition, a non-invasive evaluation of the efficacy of CNA and the incidence of syncope (MAS) and collapse (paraMAS) will take place in group 1, as well as an evaluation of the pacing percentage. After another month during the second hospitalization, the following will be performed: EPS and ECVS, and repeat CNA if ECVS does not show full parasympathetic cardiac denervation. In group 2, after 2 months, non-invasive tests will also be performed to assess and presence of MAS, paraMAS symptoms, and to assess pacing rates. After another month, during the second hospitalization, the following will be performed: EPS, ECVS and CNA. Group 1 and 2 patients will have their pacemaker set to VVI/AAI 30/min. Group 3 patients will then be evaluated for pacing rates and MAS, paraMAS symptoms. At the third visit, one month after the second invasive procedure in group 1 and 2 patients, the pacing percentage will be assessed. Patients with zero pacing percentage PM will be put on ODO/OVO/OAO-pacing off mode. Patients with a pacing percentage greater than zero PM will be set to their optimal mode. A pacing percentage of <0.1% will be treated as 0%, which will be confirmed in the ILR control. For the next 12 months, patients will be observed. During this period, at the next 4 visits repeated every 3 months, groups 1 and 2 will undergo a non-invasive assessment of CNA efficacy and bradycardia symptoms, while group 3 will be evaluated for MAS, paraMAS and pacing percentage assessment. At the 7th visit, the qualification of patients in groups 1 and 2 for discontinuation of continued pacing treatment will take place, with possible qualification for TLE.

Justification Early and late results of a new strategy which is CNA, indicate the possibility of developing an new approach that allows patients with functional bradycardia to decide whether to discontinue or optimize PM therapy. However, standardized approaches based on noninvasive and invasive techniques have not yet been validated and evaluated in a prospective, multicenter, randomized, controlled trial with long-term remote follow-up, including ILR.

DETAILED DESCRIPTION:
Visit 1- Screening, recruitment, randomization.

* ECG, PM check, NIEPS
* change the stimulation mode to DDD 50/min, AV 220ms/ VVI 50/min/ AAI 50/min
* atropine test
* laboratory tests: complete blood count, creatinine, AST, ALT, TSH, fT3, fT4, NT-proBNP, beta-HCG, K
* analysis of inclusion and exclusion criteria

Hospitalization 1-1 month from randomization Group 1- EPS, ECVS, CNA, ILR implantation Group 2- EPS, ECVS, ILR implantation Group 3- observation

Visit 2-3 months after randomization

Group 1 and 2:

* History of MAS and paraMAS symptoms and the consequences of the procedures performed.
* PM control with the assessment of the percentage of stimulation. Change settings and check PM - to assess the efficiency of own rhythm, patients will then have their pacemaker reprogrammed in DDD 50/min mode with AV 220ms or VVI 50/min. or AAI 50/min.
* ECG
* NIEPS
* 24-hour Holter ECG monitoring
* ILR control

Group 3 observation:

* History of MAS and paraMAS symptoms.
* PM control with the assessment of the percentage of stimulation.

Hospitalization 2-4 months from randomization Group 1 - EPS, ECVS, redo CNA if required Group 2 - EPS, ECVS, CNA Group 1 and 2 patients will have their pacemaker set to VVI/AAI 30/min. For patients of Groups 1 and 2 in whom the CNA proved to be ineffective, the PM will be programmed in the optimal mode for them.

Visit 3-6 months after randomization

Group 1 and 2:

* History of MAS and paraMAS symptoms and the consequences of the procedures performed.
* PM control with the evaluation of the percentage of stimulation. Changing settings and checking PM- to assess the efficiency of your own rhythm
* ECG
* NIEPS
* 24 hour Holter ECG monitoring
* ILR control Patients from groups 1 and 2, whose percentage of stimulation in PM control will be 0%, will have their PM reprogrammed to ODO/OVO/OAO - pacing off.

Group 3 observation:

* History of MAS and paraMAS symptoms.
* PM control with the assessment of the percentage of stimulation.

Visits 4, 5, 6 - consecutively 9, 12, 15 months after randomization

Groups 1 and 2:

* Anamnesis for possible symptoms of bradycardia and undesirable effects of the procedure.
* PM control
* ECG
* NIEPS
* 24-hour Holter ECG monitoring
* ILR control Patients in Groups 1 and 2 who experience symptoms of bradycardia correlated with bradycardia recorded in the ILR will resume pacing in the optimal mode for them.

During these visits, patients in Group 3 and Groups 1 and 2 who had their pacing restored/optimized will be interviewed for possible MAS and paraMAS symptoms, perform a physical examination, and check the PM with assessment of pacing percentage and pacing mode optimization.

Visit 7 - ending the study - 18 months from randomization.

Group 1 and 2:

* Anamnesis for possible symptoms of bradycardia and undesirable effects of the procedure.
* PM control
* ECG
* NIEPS
* Atropine test
* 24-hour Holter ECG monitoring
* ILR control Patients from groups 1 and 2 without symptoms of bradycardia and without asymptomatic bradycardia <40/min recorded in the ILR, after assessment by the EP-HEART TEAM (a council of two cardiologist specialists), will be qualified for the end of permanent pacing therapy. Those patients with a low risk of TLE will be qualified for TLE.

During this visit, Group 3 and Group 1 and 2 patients with previously pacing restored/optimized will be interviewed for possible MAS and paraMAS symptoms, perform a physical examination and PM check with assessment of pacing percentage and pacing mode optimisation.

The ILR will be left in place until the battery runs out or will be removed sooner at the patient's request.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pacemaker implantation before 50 years old due to sinus node and/or atrioventricular node dysfunction
* Positive response to atropine test
* Age between 18-65 years
* Signed informed consent to participate in the study

Exclusion Criteria:

* Own heart rate <30/min
* Fainting after pacemaker therapy initiation
* Persistent and sustained atrial fibrillation
* History of myocarditis
* History of myocardial infarction
* History of cardiac surgery
* History of ablation procedures
* Congenital heart defects
* Congenital atrioventricular block
* Neuromuscular and neurodegenerative diseases
* Indications for expanding the pacemaker system to ICD/CRT-D
* Pregnancy
* Renal insufficiency with GFR <30 ml/min/1.73m2
* Age below 18 and above 65 years
* HAS-BLED score >/= 3 points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoints- Composite endpoint | 18 months
  Composite endpoint including:
  * occurrence of non-traumatic loss of consciousness
  * occurrence of symptoms of presyncope state
  * determination in the loop recorder recording of events of asymptomatic bradycardia requiring permanent cardiac pacing, understood as:
    1. type II degree atrioventricular block and/or
    2. atrioventricular block of 2:1 or higher order and/or
    3. sinus bradycardia <40/min during the patient's wakefulness
    4. sinus pause >3 seconds during the patient's wakefulness
    5. cardiac pacing despite the PM setting in AAI/VVI mode 30/min after the second intervention.
Primary safety endpoints- Composite endpoint | 18 months
  Composite endpoint including:
  * death from any cause
  * peri-procedural damage to cardiac or vascular structures requiring surgical intervention not resulting in death
  * ischemic stroke not terminated by death
  * symptomatic damage to the pulmonary veins
  * symptomatic injury to the phrenic nerve
  * de-electrode device-related infective endocarditis
  * device lodge infection
  * electrode dysfunction requiring electrode replacement
  * BARC grade 2, 3 bleeding during postoperative anticoagulant therapy

SECONDARY OUTCOMES:
Secondary efficacy endpoint | 18 months
  Occurrence of non-traumatic loss of consciousness
Secondary efficacy endpoint | 18 months
  Occurrence of syncope in the course of documented bradyarrhythmia
Secondary efficacy endpoint | 18 months
  Occurrence of symptoms of pre-fainting state
Secondary efficacy endpoint | 18 months
  Occurrence of presyncope in the course of documented bradyarrhythmia
Secondary efficacy endpoint | 18 months
  Determination in the loop recorder recording of events of asymptomatic bradycardia requiring permanent pacing of the heart, understood as:
  1. atrioventricular block type II and/or
  2. atrioventricular block of 2:1 or higher order and/or
  3. sinus bradycardia <40/min during the patient's wakefulness
  4. sinus pause >3 seconds during the patient's wakefulness
  5. cardiac pacing despite the PM setting in AAI/VVI mode 30/min after the second intervention.
Secondary efficacy endpoint | 18 months
  Disabling permanent cardiac pacing at visit 3
Secondary efficacy endpoint | 18 months
  Demonstration of a statistically significant lower pacing rate in the group of patients undergoing CNA vs patients who continued PM therapy without CAN
Secondary efficacy endpoint | 18 months
  Qualification for removal of PM and TLE system
Secondary safety endpoint | 18 months
  Death from any cause
Secondary safety endpoint | 18 months
  Peri-procedural damage to cardiac or vascular structures requiring surgical intervention not resulting in death
Secondary safety endpoint | 18 months
  Ischemic stroke not terminated by death
Secondary safety endpoint | 18 months
  Symptomatic pulmonary venous injury
Secondary safety endpoint | 18 months
  Symptomatic phrenic nerve injury
Secondary safety endpoint | 18 months
  Asymptomatic phrenic nerve injury
Secondary safety endpoint | 18 months
  Electrodermal infective endocarditis
Secondary safety endpoint | 18 months
  PM implantation site infection
Secondary safety endpoint | 18 months
  Electrode dysfunction
Secondary safety endpoint | 18 months
  Occurrence of atrial tachyarrhythmias
Secondary safety endpoint | 18 months
  Development of symptoms of heart failure
Secondary safety endpoint | 18 months
  Symptoms of inadequate sinus tachycardia
Secondary safety endpoint | 18 months
  Hospitalization for any reason
Secondary safety endpoint | 18 months
  BARC grade 2, 3 bleeding during postoperative anticoagulant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw Skoczynski, PhD, Principal Investigator — 4th Military Clinical Hospital with Polyclinic, Poland; Dariusz Jagielski, PhD, Study Director — 4th Military Clinical Hospital with Polyclinic, Poland
Locations (2):
- Poland (2):
  - Mazowiecki Specialist Hospital, Radom, Masovian Voivodeship
  - Medical University of Silesia, Katowice, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Result] Rudbeck-Resdal J, Christiansen MK, Johansen JB, Nielsen JC, Bundgaard H, Jensen HK. Aetiologies and temporal trends of atrioventricular block in young patients: a 20-year nationwide study. Europace. 2019 Nov 1;21(11):1710-1716. doi: 10.1093/europace/euz206. PMID 31424500
- [Result] Chung MK, Fagerlin A, Wang PJ, Ajayi TB, Allen LA, Baykaner T, Benjamin EJ, Branda M, Cavanaugh KL, Chen LY, Crossley GH, Delaney RK, Eckhardt LL, Grady KL, Hargraves IG, True Hills M, Kalscheur MM, Kramer DB, Kunneman M, Lampert R, Langford AT, Lewis KB, Lu Y, Mandrola JM, Martinez K, Matlock DD, McCarthy SR, Montori VM, Noseworthy PA, Orland KM, Ozanne E, Passman R, Pundi K, Roden DM, Saarel EV, Schmidt MM, Sears SF, Stacey D, Stafford RS, Steinberg BA, Youn Wass S, Wright JM. Shared Decision Making in Cardiac Electrophysiology Procedures and Arrhythmia Management. Circ Arrhythm Electrophysiol. 2021 Dec;14(12):e007958. doi: 10.1161/CIRCEP.121.007958. Epub 2021 Dec 6. PMID 34865518
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Piotrowski R, Baran J, Sikorska A, Krynski T, Kulakowski P. Cardioneuroablation for Reflex Syncope: Efficacy and Effects on Autonomic Cardiac Regulation-A Prospective Randomized Trial. JACC Clin Electrophysiol. 2023 Jan;9(1):85-95. doi: 10.1016/j.jacep.2022.08.011. Epub 2022 Aug 28. PMID 36114133
- [Result] Tulecki L, Polewczyk A, Jachec W, Nowosielecka D, Tomkow K, Stefanczyk P, Kosior J, Duda K, Polewczyk M, Kutarski A. A Study of Major and Minor Complications of 1500 Transvenous Lead Extraction Procedures Performed with Optimal Safety at Two High-Volume Referral Centers. Int J Environ Res Public Health. 2021 Oct 3;18(19):10416. doi: 10.3390/ijerph181910416. PMID 34639716
- [Result] Sidhu BS, Gould J, Bunce C, Elliott M, Mehta V, Kennergren C, Butter C, Deharo JC, Kutarski A, Maggioni AP, Auricchio A, Kuck KH, Blomstrom-Lundqvist C, Bongiorni MG, Rinaldi CA; ELECTRa Investigators Group. The effect of centre volume and procedure location on major complications and mortality from transvenous lead extraction: an ESC EHRA EORP European Lead Extraction ConTRolled ELECTRa registry subanalysis. Europace. 2020 Nov 1;22(11):1718-1728. doi: 10.1093/europace/euaa131. PMID 32688392